CLINICAL TRIAL: NCT05984537
Title: A Study on the Impact of Bivalirudin Usage During Percutaneous Coronary Intervention for High-risk Plaques in the Coronary Artery on Post Percutaneous Coronary Intervention Coronary Microcirculation.
Brief Title: A Study on the Impact of Bivalirudin Usage During PCI for High-risk Plaques on Post-PCI Coronary Microcirculation.
Acronym: PCI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, ZHENG Bo, associate professor, Peking University First Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: ZHENG Bo.
Record Dates: First submitted 2023-07-23; First posted 2023-08-09 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Coronary Microvascular Dysfunction
Keywords: coronary microvascular dysfunction; computed tomography angiography; percutaneous coronary intervention; bivalirudin; heparin
MeSH Terms: interventions — bivalirudin

STUDY DESIGN:
Intervention Model Description: single-center
Who Masked: Participant
Masking Description: single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- bivalirudin group (Experimental): participants using bivalirudin during PCI
  Interventions: Drug: Bivalirudin
- standard heparin group (Active Comparator): participants using standard heparin during PCI
  Interventions: Drug: standard heparin

INTERVENTIONS:
Drug: Bivalirudin — Participants in the bivalirudin group received a one-time intravenous injection of 0.75 mg/kg during PCI, and then received a continuous intravenous infusion of 1.75 mg/kg/h for 4 hours according to the participants' condition after PCI.
  Other Names: bivalirudin anticoagulation
  Arms: bivalirudin group
Drug: standard heparin — Participants in the standard heparin group received a one-time intravenous injection of 50 U/kg of standard heparin during PCI.
  Other Names: standard heparin anticoagulation
  Arms: standard heparin group

SUMMARY:
In this study, investigators enrolled patients with coronary heart disease who were scheduled to undergo percutaneous coronary intervention (PCI) and had high-risk plaques according to computed tomography angiography (CTA). During the PCI procedure, patients will be randomly assigned to receive either bivalirudin or standard heparin anticoagulation therapy. Investigators will compare the post-PCI coronary angiography-derived index of microcirculatory resistance (CaIMR), thrombolysis in myocardial infarction (TIMI) blood flow grade, CTFC (corrected TIMI frame count), TIMI myocardial perfusion grading(TMPG), levels of troponin, and major adverse cardiac events (MACE) during a follow-up period of 6 months between the two groups. Investigators aim to explore the potential benefits of bivalirudin perioperative anticoagulation therapy in improving coronary microvascular dysfunction (CMD) after PCI for high-risk plaques in coronary artery lesions.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is one of the leading causes of death in China, with nearly 11.39 million patients affected. Percutaneous coronary intervention (PCI) is an important treatment for CAD, but despite effectively improving coronary stenosis, patients still experience the phenomenon of no-reflow (NR), which seriously affects long-term prognosis. Coronary microvascular dysfunction (CMD) during PCI is an important mechanism of NR, and previous studies have shown that immediate post-PCI CMD significantly affects long-term prognosis. Previous studies have shown that high-risk plaques identified by computed tomography angiography (CTA) before surgery in patients with stable coronary heart disease are closely related to the occurrence of NR and can serve as a predictor of NR after PCI. Therefore, CTA can identify high-risk patients for NR before PCI and has clinical value in preventing NR. Bivalirudin is a direct thrombin inhibitor that can block the continued development of blood clots. BIVAL study has shown that bivalirudin can improve post-PCI microcirculation dysfunction in patients with acute ST-segment elevation myocardial infarction, and animal experiments have shown that bivalirudin can improve thrombin-induced endothelial hyperpermeability.

In this study, investigators plan to identify high-risk coronary artery plaques early through CTA examination. Participants will be randomly assigned to receive either bivalirudin or standard heparin anticoagulation therapy. Investigators will compare the post-PCI CaIMR, thrombolysis in myocardial infarction (TIMI) blood flow grade, CTFC (corrected TIMI frame count), TIMI myocardial perfusion grading(TMPG), levels of troponin, and major adverse cardiac events (MACE) during a follow-up period of 6 months between the two groups. Investigators will also explore the possible mechanisms by which bivalirudin reduces coronary microcirculatory injury and improves endothelial function through the detection of endothelial function-related biomarkers, providing evidence for the multi-effectiveness of bivalirudin in myocardial protection.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 years or older;
2. diagnosed with non-ST-segment elevation myocardial infarction or unstable angina pectoris;
3. scheduled to undergo elective coronary angiography and intervention;
4. coronary computed tomography angiography showing high-risk plaque features within 3 months prior to the procedure;
5. voluntary participation in the study and signed informed consent.

Exclusion Criteria:

1. prior PCI of the target vessel within 3 months;
2. cardiogenic shock, active bleeding, bleeding disorders, irreversible coagulation dysfunction, severe liver dysfunction (Child-Pugh class C), severe renal dysfunction (eGFR < 30 ml/min/1.73m2), and dependence on dialysis;
3. life expectancy less than 1 year;
4. chronic total occlusion of the target vessel;
5. poor opacification of the target vessel, severe vessel overlap or distortion, and inability to completely expose the lesion site;
6. allergy to contrast agents, verapamil, or its excipients;
7. severe uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg);
8. subacute bacterial endocarditis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-04 (Estimated)

PRIMARY OUTCOMES:
CaIMR | 3 days
  The caIMR value of the target vessel immediately after PCI.
CMD | 3 days
  The proportion of target vessels with caIMR ≥ 25 and caIMR ≥ 40 immediately after PCI.

SECONDARY OUTCOMES:
clinical events | 6 months
  (1) MACE (including cardiac death, target vessel revascularization, target vessel myocardial infarction, and heart failure readmission) at 30 days and 6 months after PCI; (2) Major adverse events (including all-cause death, non-fatal myocardial infarction, unplanned revascularization, definite or probable stent thrombosis, and clinically significant bleeding events) at 30 days and 6 months.
biomarker_eNOs | 3 days
  Serum levels of eNOs after PCI.
biomarker_ET-1 | 3 days
  Serum levels of ET-1 after PCI.
biomarker_myocardial injury markers | 3 days
  Peak levels of myocardial injury markers (CK-MB and CTNI) after PCI.
imaging examination_microcirculation | 3 days
  Other indicators for assessing microcirculation during the procedure (including TMPG, TIMI frame count, and myocardial staining grade).
imaging examination_longitudinal myocardial strain | 3 days
  Changes in global longitudinal myocardial strain of the left ventricle measured by post-PCI echocardiography compared to baseline values.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Zheng, Prof, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking university first hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No